CLINICAL TRIAL: NCT04688567
Title: Patient-driven Internet Delivered Psychological Treatment in a Primary Care Context: a Randomized Controlled Trial
Brief Title: Patient-driven Internet Delivered Psychological Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr: 2019-03786
Record Dates: First submitted 2020-12-17; First posted 2020-12-30 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Anxiety Disorders and Symptoms; Internet-Based Intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The groups are predetermined based on the tool randomizer.org and blinded to the researcher assigning the participants to groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-driven iCBT (Experimental): Participants who are randomized to the experimental condition are asked to make choices regarding the structure of their treatment program
  Interventions: Behavioral: Patient-driven iCBT
- Standardized iCBT (TAU) (Active Comparator): Patients who are randomized to the control condition undergo the usual iCBT program available for anxiety disorders for a standardized time period of 8 weeks
  Interventions: Behavioral: Standardized iCBT (TAU)

INTERVENTIONS:
Behavioral: Patient-driven iCBT — 1) Participants who are randomized to the experimental condition are asked to make choices regarding the structure of their treatment by the time of the randomization call. The participant can choose which of the available treatment programs (targeting anxiety, worry, stress, sleep disorders or depression) they want to undergo, how many modules in the treatment program they want to complete and in what order, for how many weeks they want to complete the treatment as well as how much telephone contact and how much written contact they want to have with their therapist.
  Arms: Patient-driven iCBT
Behavioral: Standardized iCBT (TAU) — 2) Patients who are randomized to the control condition (standardized iCBT) undergo the usual iCBT program available for anxiety disorders for 8 weeks. The psychologist provide weekly feedback on the patient's exercises and interact with the patient via secure encrypted messages in the treatment program. A follow-up telephone call takes place at the middle of treatment and at the end of the treatment.
  Arms: Standardized iCBT (TAU)

SUMMARY:
The effect of iCBT for adults with anxiety disorders is well-known. However, drop-out rates are common. In recent years more focus has been directed to the importance of patients being active agents in their own care and to increase the patient´s involvement in health care. Studies show that involving patients´ in treatment decisions and management of their own health care can contribute to better treatment outcomes and more appropriate use of health care service.

Few studies have evaluated patient involvement in iCBT-treatment. This study aims to evaluate the effect of patient-driven iCBT-treatment for patients with anxiety disorders seeking primary care in a randomized controlled trial. The study investigates the effect of patient-driven iCBT treatment of perceptions of being able to control the treatment and on drop-out from treatment. In addition, secondary research questions investigate measures of empowerment, anxiety and depression symptoms, general disability, satisfaction with treatment and feelings of being able to cope with one's mental illness in patient-driven iCBT.

DETAILED DESCRIPTION:
The following research questions will be examined:

Primary research questions:

1. Is there a difference between participants in patient-driven digital psychological treatment, compared to standardized internet CBT, in perceptions of how much they've been able to control their treatment (measured with a questionnaire developed by the researchers for this study)?
2. What is the effect of patient-driven digital psychological treatment, compared to standardized internet CBT, on frequency of completers and completed modules among adults with anxiety disorders?

   Secondary research questions:
3. What is the effect of patient-driven digital psychological treatment, compared to standardized internet CBT, on the experience of empowerment, (measured by the "Empowerment Scale"), for adults with anxiety disorders?
4. What is the effect of patient-driven digital psychological treatment, compared to standardized internet CBT, on anxiety (measured with GAD-7), depression (measured with MADRS-S), general disability (measured with WHODAS 2.0) and steps in "valued direction" (measured with "Bull´s Eye compass") for adults with anxiety disorders?

   Associations:
5. Is there a correlation between perceptions of how much one has been able to control the treatment (measured with a questionnaire developed by the researchers for this study), feelings of being able to cope with one's mental illness (measured with Patient Enablement Instrument), how satisfied participants are with their treatment (measured vid CSQ-8), perceptions of empowerment (measured with the "Empowerment Scale") and changes in anxiety symptoms (measured with GAD-7)?
6. Does perceptions of how much participants have been affected by the pandemic of Covid-19 in their daily life correlate with anxiety symptoms (measured with GAD-7) 3 months after termination of treatment?

   Mediation:
7. What is the mediating effect of empowerment, measured by the "Empowerment Scale", on changes in anxiety symptoms (measured with GAD-7)?

ELIGIBILITY:
Inclusion Criteria:

* Has reached the age of 18
* Has access to a computer with internet connection
* Speak and understand Swedish
* Meets the diagnostic criteria for an anxiety disorder (social anxiety, GAD (Generalized Anxiety Disorder), panic disorder, obsessive-compulsive disorder or unspecified anxiety disorder)

Exclusion Criteria:

* has started medication for mental illness or made major changes regarding the medication during the past 4 weeks
* has serious suicidal thoughts or suicidal plans
* has complex comorbidity or is in need of other care for mental illness in addition to iCBT
* is receiving other psychological treatment during the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Questions of perceptions in how much one has been able to control the treatment | At the end of treatment (after 8-16 weeks depending on treatment condition)
  Perceptions in how much one has been able to control the treatment is measured by a questionnaire developed by the researchers for this study. The questionnaire consists of 9 items and each item is answered on a seven-point scale, from "Not at all" to "To a large extent".
Adherence to treatment | At the end of treatment (after 8-16 weeks depending on treatment condition)
  Adherence to treatment is measured by counting number of completed modules in the treatment program for each participant

SECONDARY OUTCOMES:
Changes in feelings of empowerment | Baseline (Pre-treatment), Middle of treatment, At the end of treatment (after 8-16 weeks depending on treatment condition) and by 3 months follow up
  Empowerment is measured with the Empowerment Scale (Rogers, Chamberlin, Ellison & Crean, 1997). The scale consists of 28 items which are answered on a four-point likert scale. Score ranges between 28 and 112. Higher scores indicates that the person feels more empowered.
Perceptions of being able to cope with one's mental illness | At the end of treatment (after 8-16 weeks depending on treatment condition) and by 3 months follow up
  Perceptions of being able to cope with one's mental illness is measured with the Patient Enablement Instrument (PEI; Howie, Heaney & Maxwell, 1997). The instrument consists of 6 items and are graded on a three-point scale. Score ranges between 0-12, with higher score indicating higher patient enablement.
Satisfaction with treatment | At the end of treatment (after 8-16 weeks depending on treatment condition) and by 3 months follow up
  Satisfaction with treatment is measured by The Client Satisfaction Questionnaire- 8 item version (CSQ-8; Attkisson & Greenfield, 1998). The questionnaire consists of 8 items and are graded on a four-point scale. Scores ranges from 8-32, with higher scores indicating higher satisfaction.
Changes in Anxiety symptoms | Baseline (Pre-treatment), Middle of treatment, At the end of treatment (after 8-16 weeks depending on treatment condition) and by 3 months follow up
  Anxiety is measured with the GAD-7 instrument (Generalized Anxiety Disorder 7 item scale). The scale consists of 7 items. The score ranges from 0 to 21, with higher scores indicating more anxiety symptoms. There are thresholds for mild, medium and severe anxiety (Spitzer, Kroenke, Williams & Löwe 2006).
Changes in Depressive symptoms | Baseline (Pre-treatment), middle of treatment, At the end of treatment (after 8-16 weeks depending on the treatment condition) and by 3 months follow up
  Symptoms of depression is measured with Madrs-s (Montgomery Åsberg Depression Rating Scale; Montgomery & Åsberg, 1979). The instrument consists of 9 items. Scores ranges from 0 to 60, with higher scores indicating more depressive symptoms. There are cut-off points for symptom severity.
Changes in General disabillity | Baseline (Pre-treatment), Middle of treatment, At the end of treatment (after 8-16 weeks depending on treatment condition) and by 3 months follow up
  General disability is measured with the 12-item version of the generic assessment tool WHO Disability Assessment Schedule (WHODAS 2.0; Rhem, Ustun, Saxena, Nelson, Chatterji, Ivis & Adlaf, 1999). Scores range from 12-60, with a higher score indicating higher disability. The instrument has established normative data.
Changes in steps towards "valued direction" | Baseline (Pre-treatment), Middle of treatment, At the end of treatment (after 8-16 weeks depending on treatment condition) and by 3 months follow up
  Steps towards "valued direction" is measured with "the Bull´s Eye Values Survey" (Lundgren, Louma, Dahl, Strohsal & Melin, 2012).
10. Questions about how much one has been affected by the pandemic of Covid-19 | By 3 months follow up
  Perceptions about how much one has been affected by the pandemic of Covid-19 is measured by a questionnaire developed by the researchers for this study. The questionnaire consists of 7 items that is answered on a seven-point scale. 1 indicating= To a very large extent for the worse; 4= not at all / not relevant; 7= to a very large extent for the better.

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Nissling, Phd-student, Principal Investigator — Department of Psychology, University of Gothenburg, Sweden; Martin Kraepelien, PhD, Study Director — Centre for Psychiatry Research, Department of Clinical Neuroscience, Karolinska Institutet, Sweden; Viktor Kaldo, Professor, Study Director — Centre for Psychiatry Research, Department of Clinical Neuroscience, Karolinska Institutet, Sweden; Dominique Hange, Docent, Study Director — General Medicine, School of Public Health and Community Medicine, Sahlgrenska Academy, Sweden; Anna Larsson, Psy M, Study Director — Research, Development, Education and Innovation, Primary Health Care, Region Västra Götaland,Sweden; Sandra Weineland, Docent, Principal Investigator — Department of Psychology, University of Gothenburg, Sweden
Locations (1):
- Department of Psychology, University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We will share the data if a corresponding author or otherwise authorized person asks for it
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Nissling L, Kraepelien M, Kaldo V, Hange D, Larsson A, Persson M, Weineland S. Effects of patient-driven iCBT for anxiety in routine primary care and the relation between increased experience of empowerment and outcome: A randomized controlled trial. Internet Interv. 2021 Sep 21;26:100456. doi: 10.1016/j.invent.2021.100456. eCollection 2021 Dec. PMID 34603972